CLINICAL TRIAL: NCT04643288
Title: Clinical and Radiographic Evaluation of Open Flap Debridement With or Without Nanocrystalline Hydroxyapatite Bone Graft in Management of Periodontal Intrabony Defects
Brief Title: Nanocrystalline Hydroxyapatite Bone Substitute for Treating Periodontal Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weam Ahmed Elbattawy (Other)
Responsible Party: Sponsor-Investigator, Weam Ahmed Elbattawy, Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: nano version 1
Record Dates: First submitted 2020-11-14; First posted 2020-11-25 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Chronic Periodontitis
Keywords: periodontal intrabony defects
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OFD control group (Experimental): open flap debridement for periodontal intrabony defects
  Interventions: Procedure: open flap debridement
- n-HA bone graft intervention group (Experimental): Nanocrystalline Hydroxyapatite (n-HA) bone graft substitute was added to periodontal intrabony defects
  Interventions: Procedure: open flap debridement; Procedure: n-HA bone graft

INTERVENTIONS:
Procedure: open flap debridement — open flap debridement for managing two and three walls intrabony periodontal defects
Procedure: n-HA bone graft — Nanocrystalline Hydroxyapatite bone graft substitute for managing two and three walls intrabony periodontal defects
  Arms: n-HA bone graft intervention group

SUMMARY:
The present clinical trial included 20 patients (11 females and 9 males, aged 36 to 56 years) suffering from moderate or advanced chronic periodontitis. Subjects were recruited from the outpatient clinic, Department of Oral Medicine and Periodontology, Faculty of Dentistry, Cairo University. This clinical trial was meant to assess clinically and radiographically the possible predictable results regarding the use of nanocrystalline hydroxyapatite bone graft substitute together with open flap debridement versus open flap debridement alone in the treatment of periodontal intrabony defects.

DETAILED DESCRIPTION:
periodontal intrabony defects in patients with moderate or advanced chronic periodontitis were treated with open flap debridement only in the control group while open flap debridement and Nanocrystalline Hydroxyapatite bone graft substitute was performed for the intervention group. probing pocket depth, clinical attachment level, gingival index, plaque index, gingival recession and bone defect area were assessed at baseline and six months post surgically to evaluate the possible improvement in the clinical and radiographic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients
* diagnosed with moderate to advanced chronic periodontitis
* periodontal defects with at least one site with probing pocket depth (PPD) ≥ 5mm, clinical attachment loss (CAL) ≥ 4mm and two or three-walled intra-bony defects ≥ 3mm
* evidence of intrabony defects using periapical radiographs

Exclusion Criteria:

* teeth with suprabony defects or 1-wall intrabony defects
* pregnant or lactating women
* patients taking any medication 3 months prior to the study
* patients receiving any periodontal treatment 6 months prior to study initiation
* former or current smokers.

Ages: 35 Years to 56 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
change in probing pocket depth | baseline and after six months
  William's graduated periodontal probe used to measure probing pocket depth from the gingival margin to the base of the sulcus

SECONDARY OUTCOMES:
change in clinical attachment level | baseline and after six months
  William's graduated periodontal probe used to measure clinical attachment level from the cementoenamel junction to the base of the sulcus
change in the bone defect area | baseline and after six months
  periodical digital radiographs using Digora software to measure the bone defect area

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt